CLINICAL TRIAL: NCT02190045
Title: Wii-Fit For Balance And Gait In Elderly Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Arkansas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kalpana Padala, MD, Staff Physician, Central Arkansas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 404039
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-01

CONDITIONS: Gait, Unsteady; Postural Balance
Keywords: Balance; gait; Wii-Fit
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wii-Fit program (Experimental): Wii-Fit exercises will be adminstered for 45 minutes 3 days a week for 8 weeks
  Interventions: Other: Wii-Fit exercises
- Cognitive remediation program (Placebo Comparator): Cognitive remediation exercises will be adminstered for 45 minutes 3 days a week for 8 weeks
  Interventions: Other: Cognitive remediation exercises

INTERVENTIONS:
Other: Wii-Fit exercises — Wii-Fit exercises will be administered for 45 minutes 3 days of the week for 8 weeks
  Arms: Wii-Fit program
Other: Cognitive remediation exercises — Cognitive Remediation exercises will be administered for 45 minutes 3 days of the week for 8 weeks
  Arms: Cognitive remediation program

SUMMARY:
Falls are a major public health problem. They are the leading cause of injuries and injury-related deaths in those aged over 65 years. Balance and gait abnormalities are major reasons for falls in elderly. Exercise interventions improve gait and balance in the elderly. Despite the many proven benefits of exercise, many older adults in the US remain sedentary. This study targets at improving balance and gait with use of Wii-Fit as an exercise program.

DETAILED DESCRIPTION:
Objectives/Rationale Falls are a major public health problem. They are the leading cause of injuries and injury-related deaths in those aged over 65 years. Balance and gait abnormalities are major reasons for falls in elderly. Exercise interventions improve gait and balance in the elderly. Despite the many proven benefits of exercise, many older adults in the US remain sedentary. This study targets at improving balance and gait with use of Wii-Fit as an exercise program.

Specific aims

1. To establish the safety, feasibility, and efficacy of an 8-week Wii-Fit program to improve measures of balance, and gait in older adults, compared to a cognitive remediation program, Brain fitness.
2. To compare the effect of an 8-week Wii-Fit program to Brain fitness program, on measures of biomechanical assessment, adherence, safety, physical activity, fear of fall, enjoyment, functional status, cognition and quality of life.

Design 8-week, randomized, parallel group, active intervention study Methods Patients will be recruited via IRB approved flyers posted in various locations of the Little Rock and North Little Rock CAVHS campuses and via referrals from the CAVHS providers. Thirty elderly Veterans will be randomly assigned to Wii-Fit arm or Brain fitness arm. Both groups will participate in the intervention for approximately 45 minutes 3 days a week for 8 weeks. Outcome measures will be assessed at baseline, and approximately week 4 and after completion of week 8. Balance and gait will be assessed by Berg Balance Scale. Secondary outcome measures include biomechanical testing for gait and balance, Safety, Adherence, measures of functional status, cognition, quality of life, fear of falling, physical activity and physical activity enjoyment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 60 years
* Fall risk as measured by Berg Balance Scale (BBS) is ≤ 52
* Normal cognition as measured by Mini Mental State Exam (MMSE ≥ 24)
* Able to consent

Exclusion Criteria:

* Subjects using wheel chair or walkers for mobility
* Subjects with absolute contraindications per ACSM guidelines
* Any medical condition (per the relative contraindications per ACSM guidelines below) that in the opinion of the study physician is likely to compromise their ability to safely participate in the exercise program.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpana Padala, MD, Principal Investigator — Central Arkansas Veterans Healthcare System
Locations (1):
- Central Arkansas Veterans Healthcare System (3J/NLR), North Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Padala KP, Padala PR, Lensing SY, Dennis RA, Bopp MM, Parkes CM, Garrison MK, Dubbert PM, Roberson PK, Sullivan DH. Efficacy of Wii-Fit on Static and Dynamic Balance in Community Dwelling Older Veterans: A Randomized Controlled Pilot Trial. J Aging Res. 2017;2017:4653635. doi: 10.1155/2017/4653635. Epub 2017 Feb 5. PMID 28261500

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wii-Fit Program | Cognitive Remediation Program
Started | 15 | 15
Completed | 12 | 15
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wii-Fit Program | Cognitive Remediation Program | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (8.1) | 69.0 (3.8) | 68.0 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 13 | 13 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Non-Hispanic Caucasian | 8 | 12 | 20
  Race: Non-Hispanic African American | 7 | 3 | 10
Berg Balance Scale [Mean (Standard Deviation); unit: units on a scale] | 48.5 (2.6) | 50.1 (2.5) | 49.3 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale
Description: The primary efficacy outcome was the Berg Balance Scale (BBS), which assesses balance impairments in older adults and is a good measure of static and dynamic stability. It consists of 14 tasks performed in a standardized order with each task scored on a five-point scale according to quality or time ranging from "0" (lowest level of function) to "4" (highest level). The maximum score is 56. BBS has an excellent inter-rater reliability (0.98). A change of four points is considered the minimally detectable change for community dwelling older adults that ambulate without an assistive device.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wii-Fit Program | Cognitive Remediation Program
Number analyzed (Participants) | 15 | 15
units on a scale | 48.5 (2.6) | 50.1 (2.5)

2. Secondary Outcome: Quality of Life (SF-36)
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Functional Status Measures
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Activities Specific Balance Confidence Scale
Time Frame: 8 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Modified Mini- Mental Exam
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Wii-Fit Program | Cognitive Remediation Program
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes